CLINICAL TRIAL: NCT00374504
Title: Prediction of Postoperative Pain by an Electrical Pain Stimulus
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: 01 2745584
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-02

CONDITIONS: Cesarean Section

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The aim of this study is to evaluate a possible correlation between predictive precesarean section pain and development of postcaesarean section pain using the PM.

Patients and Methods 46 healthy pregnant women scheduled for elective cesarean section is included after informed consent. The standard operation procedures included spinal anesthesia, paracetamol 1 g 8 hourly, diclofenac 50 mg 8 hourly and oxycontine 10 mg x 2. Morphine was used for break-through pain.

Before cesarian section the threshold for sensory and pain were measured 3 times, and the average was used for analyses. After cesarian section a blinded midwife assess the pain at rest and during mobilization every 12th hours over 2 days score.

Data was analyzed using AUC and non-parametric test, P < 0,05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women scheduled for elective cesarean section

Exclusion Criteria:

* ASA III -IV
* Chronic pain conditions.
* Pacemaker.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46

CONTACTS AND LOCATIONS:
Overall Officials: Per Rotbøll Nielsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital, Rrigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Nielsen PR, Norgaard L, Rasmussen LS, Kehlet H. Prediction of post-operative pain by an electrical pain stimulus. Acta Anaesthesiol Scand. 2007 May;51(5):582-6. doi: 10.1111/j.1399-6576.2007.01271.x. PMID 17430320